CLINICAL TRIAL: NCT01632228
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Study Evaluating the Efficacy and Safety of Onartuzumab in Combination With Bevacizumab or Onartuzumab Monotherapy in Patients With Recurrent Glioblastoma
Brief Title: A Study of Onartuzumab (MetMAb) in Combination With Bevacizumab Compared to Bevacizumab Alone or Onartuzumab Monotherapy in Participants With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27819; 2011-005912-27 (EudraCT Number)
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; onartuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Onartuzumab + Bevacizumab (Experimental): All participants will receive onartuzumab intravenous (IV) infusion followed by bevacizumab IV infusion every 3 weeks.
  Interventions: Drug: Bevacizumab; Drug: Onartuzumab
- Placebo + Bevacizumab (Active Comparator): All participants will receive placebo matched with onartuzumab followed by bevacizumab IV infusion every 3 weeks.
  Interventions: Drug: Bevacizumab; Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab — Participants will receive bevacizumab 15 milligrams per kilogram (mg/kg) IV infusion every 3 weeks until disease progression, unacceptable toxicity, participants or physician decision to discontinue, or death.
Drug: Onartuzumab — Participants will receive onartuzumab 15 mg/kg IV infusion every 3 weeks until disease progression, unacceptable toxicity, participants or physician decision to discontinue, or death.
  Other Names: MetMAb, RO5490258
  Arms: Onartuzumab + Bevacizumab
Drug: Placebo — Participants will receive placebo matched with onartuzumab until disease progression, unacceptable toxicity, participants or physician decision to discontinue, or death.
  Arms: Placebo + Bevacizumab

SUMMARY:
This randomized, double-blind, placebo-controlled, multicenter phase II study will evaluate the safety and efficacy of onartuzumab in combination with bevacizumab as compared to bevacizumab alone in participants with recurrent glioblastoma. Participants will be randomized 1:1 to receive either placebo plus bevacizumab every 3 weeks, or onartuzumab plus bevacizumab. Study treatment will continue until disease progression, unacceptable toxicity, participants or physician decision to discontinue, or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma at first recurrence after concurrent or adjuvant chemoradiotherapy
* Imaging confirmation of first tumor progression or regrowth as defined by RANO criteria
* Prior treatment with temozolomide
* No more than one prior line of chemotherapy
* No prior treatment with bevacizumab or other vascular endothelial growth factor (VEGF)- or VEGF-receptor-targeted agent
* No prior exposure to experimental treatment targeting either hepatocyte growth factor (HGF) or Met pathway
* No prior treatment with prolifeprospan 20 with carmustine wafer
* No prior intracerebral agent
* Recovery from the toxic effects of prior therapy
* No evidence of recent hemorrhage on baseline magnetic resonance imaging (MRI) of the brain
* No need for urgent palliative intervention for primary disease (e.g. impending herniation)
* Karnofsky performance status greater than or equal to (>=) 70 percent (%)
* Stable or decreasing dose of corticosteroids within 5 days prior to randomization
* Prior therapy with gamma knife or other focal high-dose radiotherapy is allowed, but the participant must have subsequent histologic documentation of recurrence, unless the recurrence is a new lesion outside the irradiated field
* Participants who have undergone recent surgery for recurrent or progressive tumor are eligible provided that: surgery must have confirmed the recurrence, a minimum of 28 days must have elapsed from the day of surgery to randomization and for core or needle biopsy, a minimum of 7 days must have elapsed prior to randomization, and craniotomy or intracranial biopsy site must be adequately healed and free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of randomization
* Availability of formalin fixed paraffin embedded tumor tissue representative of glioblastoma

Exclusion Criteria:

* Pregnant or lactating women
* Inadequate hematologic, renal or liver function
* History or presence of serious cardio-vascular disease
* New York Heart Association Grade II or greater congestive heart failure
* History of another malignancy in the previous 3 years, except for in situ cancer or basal or squamous cell skin cancer
* Inadequately controlled hypertension (defined as systolic blood pressure greater than [>]150 millimeter of mercury (mmHg) and/or diastolic blood pressure >100 mmHg while on antihypertensive medication)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Known hypersensitivity to any excipients of onartuzumab or bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2016-01-21 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as Assessed by Investigator According to Response Assessment in Neuro-Oncology (RANO) Criteria | Baseline until disease progression, intolerable toxicity, participant or physician decision, or death, whichever occurs first (assessed every 6 weeks up to 18 months)
Progression-free survival (PFS) as Assessed by Investigator According to RANO Criteria (in Participants With Met-Positive Glioblastoma) | Baseline until disease progression, intolerable toxicity, participant or physician decision, or death, whichever occurs first (assessed every 6 weeks up to 18 months)

SECONDARY OUTCOMES:
Overall Survival (All Participants) | Baseline until death (up to approximately 18 months)
Percentage of Participants who Survived at Month 9 (All Participants) | Month 9
Percentage of Participants who are Progression Free at Month 6, as Assessed by RANO Criteria (All Participants) | Month 6
Percentage of Participants With Objective Response (OR), as Assessed by RANO Criteria (All Participants) | Baseline until disease progression, intolerable toxicity, participant or physician decision, or death, whichever occurs first (assessed every 6 weeks up to 18 months)
Duration of Response, as Assessed by RANO Criteria | Baseline until disease progression, intolerable toxicity, participant or physician decision, or death, whichever occurs first (assessed every 6 weeks up to 18 months)
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to approximately 3 years 8 months
Percentage of Participants With Serum Anti-Therapeutic Antibody (ATAs) to Onartuzumab | Predose (0 hour) on Day 1 of Cycles 1, 2, 3, 4, at study completion or study drug discontinuation visit (up to approximately 3.5 years; Cycle length: 21 days)
Overall Survival (in Participants With Met-Positive Glioblastoma) | Baseline until death (up to approximately 18 months)
Percentage of Participants who Survived at Month 9 (in Participants With Met-Positive Glioblastoma) | Month 9
Percentage of Participants who are Progression Free at Month 6, as Assessed by RANO Criteria (in Participants With Met-Positive Glioblastoma) | Month 6
Percentage of Participants With Objective Response (OR), as Assessed by RANO Criteria (in Participants With Met-Positive Glioblastoma) | Baseline until disease progression, intolerable toxicity, participant or physician decision, or death, whichever occurs first (assessed every 6 weeks up to 18 months)
Duration of Response, as Assessed by RANO Criteria (in Participants With Met-Positive Glioblastoma) | Baseline until disease progression, intolerable toxicity, participant or physician decision, or death, whichever occurs first (assessed every 6 weeks up to 18 months)
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in Participants With Met-Positive Glioblastoma | Baseline up to approximately 3 years 8 months
Minimum Observed Serum Concentration (Cmin) of Onartuzumab | predose (0 hour) on Day 1 of Cycles 1, 2, 3, 4, at study completion or study drug discontinuation visit (up to approximately 3.5 years) (Cycle length: 21 days; infusion duration: Onartuzumab 60 minutes)
Maximum Observed Serum Concentration (Cmax) of Onartuzumab | predose (0 hour) and 30 minutes post dose on Day 1 of Cycles 1, 2, 3, 4, at study completion or study drug discontinuation visit (up to approximately 3.5 years) (Cycle length: 21 days; infusion duration: Onartuzumab 60 minutes)
Minimum Observed Serum Concentration (Cmin) of Bevacizumab | predose (0 hour) on Day 1 of Cycles 1, 2, 3, 4, at study completion or study drug discontinuation visit (up to approximately 3.5 years) (Cycle length: 21 days; infusion duration: Bevacizumab 90 minutes)
Maximum Observed Serum Concentration (Cmax) of Bevacizumab | predose (0 hour) and 30 minutes post dose on Day 1 of Cycles 1, 2, 3, 4, at study completion or study drug discontinuation visit (up to approximately 3.5 years) (Cycle length: 21 days; infusion duration: Bevacizumab 90 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (19):
  - University of Alabama At Birmingham; Neuro-Oncology, Birmingham, Alabama
  - Cedars Sinai Medical Center; Neurosurgery, Los Angeles, California
  - UCLA, Los Angeles, California
  - USCF - Neurosurgery, San Francisco, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Florida Cancer Specialists - Englewood, Englewood, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - North Western Univ; Neurology, Chicago, Illinois
  - Northshore University Health System; Cardiology, Evanston, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Hatton Research Institutes, Cincinnati, Ohio
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Baylor Research Inst., Dallas, Texas
  - University of Virgina, Charlottesville, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Seattle Cancer Care Alliance; Investigational Drug Service, Seattle, Washington
- Canada (6):
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Princess Margaret Hospital; Pencer Brain Tumour Centre, 18-727, Toronto, Ontario
  - McGill University; Montreal Neurological Institute; Oncology, Montreal, Quebec
  - CHUS Hopital Fleurimont; CRC, Sherbrooke, Quebec
- France (9):
  - Hopital Avicenne; Neurologie, Bobigny
  - Hopital neurologique Pierre Wertheimer - CHU Lyon; Neurologie, Bron
  - Hopital Roger Salengro, Lille
  - Hopital de La Timone - CHU de Marseille; Service de neuro-oncologie - Hôpital Adultes - 12ème étage, Marseille
  - Centre Val Aurelle Paul Lamarque; Medecine B3, Montpellier
  - Hôpital Central; Departement de Neuro-Oncologie, Nancy
  - Hopital Pitié Salpétrière - CHU; Service de neurologie 2 - Mazarin, Paris
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Hopital Purpan, Toulouse
- Germany (8):
  - Universitätsklinikum Bonn; Medizinische Klinik und Poliklinik I; Allgemeine Innere Medizin, Bonn
  - Universitätsklinikum Köln, Cologne
  - Klinikum Joh.Wolfg.Goethe-UNI Senckenbergisches Institut für Neuroonkologie, Frankfurt am Main
  - Universitatsklinikum Hamburg-Eppendorf; Klinik und Poliklinik fur Neurochirurgie, Hamburg
  - Ärztehaus Velen, Ibbenbühren
  - Klinikum der Johannes Gutenberg Uni Mainz; Studienz. Neurologie, Klinik und Poliklinik Neurologie, Mainz
  - Uni Klinikum München - Großhardern; Med. Klinik U. Poliklinik III - Abt. Onkologie u. Hämatologie, München
  - Pius-Hospital, Oldenburg
- Italy (8):
  - Ospedale Bellaria; U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - Presidio Ospedaliero Marconi Bufalini; U.O. di Oncologia, Cesena, Emilia-Romagna
  - A.O. Universitaria Di Parma; Oncologia Medica, Parma, Emilia-Romagna
  - Spedali Civili di Brescia, Brescia, Lombardy
  - Fondazione IRCCS Ospedale Maggiore Policlinico; Gastroenterologia, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico C. Besta; Neuro-oncologia Sperimentale e Terapia Genica, Milan, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Az. Osp. Pisana Ospedale S. Chiara; U.O. Di Reumatologia, Pisa, Tuscany
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Clinic i Provincial; Servicio de Farmacia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
- Switzerland (2):
  - HUG; Oncologie, Geneva
  - Universitätsspital Zürich; Klinik für Neurologie, Zurich
- United Kingdom (3):
  - Bristol Haematology and Oncology Centre, Bristol
  - Sarah Cannon Research Institute, London
  - Nottingham City Hospital; David Evans Centre, Nottingham